CLINICAL TRIAL: NCT02101515
Title: Randomized Control Trial of Usual Labor Versus Extended Second Stage
Brief Title: Randomized Control Trial of Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, alexis gimovsky, Fellow in Maternal Fetal Medicine, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13D.590
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-01

CONDITIONS: Labor Complications
Keywords: randomized controlled trial; labor complications; cesarean section; second stage
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Labor (Placebo Comparator): Immediate delivery after 3 hours with epidural or 2 hours without epidural
  Interventions: Other: Length of Second Stage
- Extended (Experimental): Immediate delivery after 4 hours with an epidural or 3 hours without an epidural
  Intervention: one additional hour for the second stage of labor
  Length of second stage in extended arm is 3 hours without epidural and 4 hours with epidural.
  Interventions: Other: Length of Second Stage

INTERVENTIONS:
Other: Length of Second Stage — The experimental group will have one additional hour in the second stage of labor

SUMMARY:
The hypothesis of this study is that extending the second stage of labor beyond current American College of Obstetricians and Gynecologists suggestions can reduce the cesarean delivery rate. The cesarean delivery rate in the United States is around 30 percent. This is a number that continues to be increasing over the last few decades and will continue to climb. Each subsequent cesarean section puts the mother and baby at increased risk for postpartum hemorrhage, bowel and bladder injury, abnormal placentation, febrile morbidity and death. The most common reason for a cesarean delivery is a repeat cesarean delivery. One way to reduce this number is to prevent the first cesarean delivery. The aim of this study is evaluate if extending the second stage of labor affects the cesarean delivery rate and subsequent perinatal morbidity.

DETAILED DESCRIPTION:
1. Consent at the time of admission or in the office
2. 2nd stage starts at full dilation
3. Randomization occurs at 2 hours without epidural or 3 hours with epidural, stratified by epidural status
4. Randomization scheme is according to a predetermined computer-generated block randomization scheme with block sizes of 6,8 and12 (random blocks).
5. Sequentially numbered and sealed opaque envelopes prepared according to the randomization scheme and delivered to a secure container in labor and delivery suite to maintain concealed treatment allocation.
6. At the 3 hour mark, the next number envelope is pulled and opened by the physician/nurse to reveal the designated group. At this point the patient is considered randomized.
7. Provider preference for cesarean delivery, operative vaginal delivery, continued pushing, with intention-to-treat analysis
8. Those that require cesarean delivery - usual perioperative management
9. Early termination criteria: emergency cesarean delivery, category 3 fetal heart tracing

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* singleton pregnancies
* cephalic presentation
* 36.0-41.6 weeks
* age 18 and older

Exclusion Criteria:

* Category 3 fetal heart tracing
* major congenital anomalies
* multiples
* planned cesarean delivery
* intrauterine fetal demise
* Trial of labor after cesarean

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Gimovsky, MD, Principal Investigator — Thomas Jefferson University; Vincenzo Berghella, MD, Study Chair — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hosptial, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Please contact Dr. Gimovsky at agimovsky@mfa.gwu.edu

REFERENCES:
- [Derived] Gimovsky AC, Phillips JM, Amero M, Levine J, Berghella V. Prolonged second stage effect on pelvic floor dysfunction: a follow up survey to a randomized controlled trial. J Matern Fetal Neonatal Med. 2022 Dec;35(25):5520-5525. doi: 10.1080/14767058.2021.1887122. Epub 2021 Feb 14. PMID 33586572
- [Derived] Gimovsky AC, Berghella V. Randomized controlled trial of prolonged second stage: extending the time limit vs usual guidelines. Am J Obstet Gynecol. 2016 Mar;214(3):361.e1-6. doi: 10.1016/j.ajog.2015.12.042. PMID 26928148

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Labor: Immediate delivery after 3 hours with epidural or 2 hours without epidural
  Length of Second Stage: The experimental group will have one additional hour in the second stage of labor
  n = 37
- Extended: Immediate delivery after 4 hours with an epidural or 3 hours without an epidural
  Intervention: one additional hour for the second stage of labor
  Length of second stage in extended arm is 3 hours without epidural and 4 hours with epidural.
  Length of Second Stage: The experimental group will have one additional hour in the second stage of labor
  n = 41
Period: Overall Study
Arm/Group | Usual Labor | Extended
Started | 37 | 41
Completed | 37 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Labor | Extended | Total
Number analyzed (Participants) | 37 | 41 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (5.4) | 27.6 (4.7) | 28.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 11 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 11 | 20
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Epidural anesthesia [Number; unit: participants] | 37 | 41 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Delivered by Cesarean
Description: Number of patients delivered by cesarean delivery for the extended labor group
Time Frame: At time of delivery, up to 4 hours of the second stage for "Extended group" and 3 hours for "Usual group"
Measure: Count of Participants; unit: Participants
Groups:
- Extended: Immediate delivery after 4 hours with an epidural or 3 hours without an epidural
  Intervention: one additional hour for the second stage of labor
  Length of second stage in extended arm is 3 hours without epidural and 4 hours with epidural.
  Length of Second Stage: The experimental group will have one additional hour in the second stage of labor
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 16 | 8
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 0.45, 95% CI 2-sided [0.22 to 0.93]

2. Secondary Outcome: Number of Newborns With Umbilical Artery pH < 7.10
Description: Umbilical artery pH is a marker for adverse neurological outcomes. Umbilical artery pH <7.10 has been proposed as a threshold for identifying fetuses who might develop pathologic fetal acidosis and fetal injury.
Time Frame: at time of delivery, 4 hours second stage for "Extended" 3 hours second stage for "Usual"
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 0 | 0

3. Secondary Outcome: Postpartum Hemorrhage
Description: Number of participants who experienced a postpartum hemorrhage
Time Frame: at time of delivery, 4 hours second stage for "Extended" 3 hours second stage for "Usual"
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 3 | 8
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 2.41, 95% CI 2-sided [0.67 to 8.40]

4. Other Pre Specified Outcome: Operative Vaginal Delivery
Time Frame: at time of delivery, 4 hours second stage for "Extended" 3 hours second stage for "Usual"
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 14 | 12
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.41 to 1.45]

5. Other Pre Specified Outcome: Spontaneous Vaginal Delivery
Time Frame: at time of delivery, 4 hours second stage for "Extended" 3 hours second stage for "Usual"
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 7 | 21
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 2.71, 95% CI 2-sided [1.30 to 5.62]

6. Other Pre Specified Outcome: Endometritis
Description: Clinical diagnosis of postpartum endometritis of the mother
Time Frame: at time of delivery until maternal discharge, usually < 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 1 | 1
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.06 to 13.92]

7. Other Pre Specified Outcome: Transfusion
Description: Any transfusion of packed red blood cells to the mother or any other blood products given.
Time Frame: at time of delivery until maternal discharge, usually < 5 days
Measure: Number; unit: participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
participants | 0 | 1

8. Other Pre Specified Outcome: 3rd/4th Degree Laceration
Description: 3rd or 4th degree laceration or cervical laceration diagnosed at delivery
  Third degree lacerations extend through the fascia and musculature of the perineal body and involve some or all of the fibers of the external anal sphincter (EAS) and/or the internal anal sphincter.
  Third degree lacerations are subclassified as follows:
  * 3a: <50 percent of EAS thickness is torn
  * 3b: >50 percent of EAS thickness is torn
  * 3c: IAS is torn (in addition to complete rupture of the EAS)
    * Fourth degree lacerations involve the perineal structures, EAS, IAS, and the rectal mucosa.
Time Frame: at time of delivery, 4 hours second stage for "Extended" 3 hours second stage for "Usual"
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 1 | 6
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 5.41, 95% CI 2-sided [0.68 to 42.90]

9. Other Pre Specified Outcome: Number of Participants With Shoulder Dystocia
Time Frame: at time of delivery, 4 hours second stage for "Extended" 3 hours second stage for "Usual"
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 0 | 1

10. Other Pre Specified Outcome: Neonatal Intensive Care Unit Admission (Neonates)
Description: One neonate was analyzed per mother
Time Frame: Birth until neonatal discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 14 | 13
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 0.8, 95% CI 2-sided [0.46 to 1.54]

11. Other Pre Specified Outcome: Chorioamnionitis
Description: Clinical diagnosis of Chorioamnionitis of the mother
Time Frame: at time of delivery, 4 hours second stage for "Extended" 3 hours second stage for "Usual"
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 13 | 11
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.39 to 1.49]

12. Other Pre Specified Outcome: Neonatal Sepsis (Neonate)
Description: Diagnosed by neonatology, one neonate was analyzed per mother
Time Frame: until neonatal discharge, usually < 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 0 | 0

13. Other Pre Specified Outcome: Birth Weight (Neonate)
Description: One neonate was analyzed per mother
Time Frame: at time of delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
grams | 3506 (534) | 3437 (527)
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; p = 0.6, t-test, 2 sided

14. Other Pre Specified Outcome: Neonatal Seizures (Neonate)
Description: Diagnosed by neonatology, one neonate was analyzed per mother
Time Frame: until discharge, usually < 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 0 | 0

15. Other Pre Specified Outcome: Neonatal Length of Stay (Neonate)
Description: one neonate was analyzed per mother
Time Frame: until neonatal discharge, usually < 5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
days | 4.03 (5.64) | 2.66 (1.02)

16. Other Pre Specified Outcome: Neonatal Mortality (Neonate)
Description: one neonate was analyzed per mother
Time Frame: early neonatal mortality (within 7 days of birth).
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 0 | 0

17. Other Pre Specified Outcome: Continuous Positive Airway Pressure or Greater (Neonate) Such as Intubation, Mechanical Ventilation, Nasal Intermittent Positive Pressure Ventilation, High-frequency Oscillatory Ventilation
Description: Number of neonates who required continuous positive airway pressure or greater.
Time Frame: Until neonatal discharge, usually < 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Labor | Extended
Number analyzed (Participants) | 37 | 41
Participants | 3 | 1
Statistical Analysis 1: Comparison: Extended; Test type: Superiority or Other; Risk Ratio (RR) = .3, 95% CI 2-sided [0.03 to 2.77]

ADVERSE EVENTS:
Arm/Group | Usual Labor | Extended
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/41
Other Adverse Events (participants affected / at risk) | 0/37 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes